CLINICAL TRIAL: NCT03825016
Title: Lidocaine Infusion Versus Oral Diclofenac During Outpatient Hystroscopy: A Randomized Clinical Trial
Brief Title: Lidocaine Infusion in Hystroscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed S Sweed, MD, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AS1855
Record Dates: First submitted 2019-01-30; First posted 2019-01-31 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Lidocaine; Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine (Experimental): Lidocaine Hydrochloride
  Interventions: Drug: Lidocaine Hydrochloride
- Diclofenac (Experimental): Oral Diclofenac
  Interventions: Drug: Diclofenac Sodium

INTERVENTIONS:
Drug: Lidocaine Hydrochloride — Lidocaine infusion on hystroscopic media during office hystroscopy
  Arms: Lidocaine
Drug: Diclofenac Sodium — Oral Diclofenac Sodium
  Arms: Diclofenac

SUMMARY:
Lidocaine infusion in hystroscopic media versus oral diclofenac

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35 years
* BMI 18.5-30 kg/m2
* Diagnostic hystroscope

Exclusion Criteria:

* Previous cervical surgery
* Cervical stenosis
* PID
* allergy to NSAID
* Gastritis or peptic ulcer

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Degree of pain "measured by visual analogue scale" | 1 hour
  measured by visual analogue scale

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt